CLINICAL TRIAL: NCT06593756
Title: Validation of Techniques for Hemodynamic Monitoring and Prediction of Fluid Responsiveness in Patients Undergoing Venoarterial Extracorporeal Membrane Oxygenation - A Prospective Diagnostic Accuracy Study ("HemodynamECMOnitoring-VA Study")
Brief Title: Hemodynamic Monitoring and Fluid Responsiveness in Venoarterial Extracorporeal Membrane Oxygenation (VA ECMO) - "HemodynamECMOnitoring-VA Study"
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Thomas Staudinger, Univ.-Prof. Dr., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1613/2023
Record Dates: First submitted 2024-05-03; First posted 2024-09-19 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: ECMO Treatment; ARDS; Pneumonia; Intensive Care; Hemodynamic Monitoring; Fluid Responsiveness
Keywords: VV ECMO; Extracorporeal Membrane Oxygenation; ARDS; Intensive Care Medicine; Critical Care Medicine; Hemodynamic Monitoring; Fluid Responsiveness; Passive Leg Raising; Pulse Contour Analysis; Transpulmonary Thermodilution; Bioreactance; Pulse Pressure Variation; End-expiratory Occlusion Test; End-inspiratory Occlusion Test; Cardiac Output; LVOT VTI; Stroke Volume; Vena Cava Ultrasound
MeSH Terms: conditions — Pneumonia | interventions — Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Entire Study Population (Experimental): The entire study population will undergo serial hemodynamic assessments throughout the course of ECMO therapy. Hemodynamic variables are obtained using transthoracic echocardiography, uncalibrated pulse contour analysis, and optionally - depending on device availability - transpulmonary thermodilution, bioreactance and esophageal doppler. Maneuvers for assessing volume responsiveness include passive leg raising (PLR), respiratory pulse pressure variation (PPV), stroke volume variation (SVV), inferior vena cava ultrasound (IVC), and end-inspiratory or end-expiratory occlusion tests.
  Interventions: Device: Transthoracic Echocardiography; Device: Uncalibrated Pulse Contour Analysis; Device: Transpulmonary Thermodilution/Calibrated Pulse Contour Analysis; Device: Esophageal Doppler; Device: Bioreactance; Diagnostic Test: Passive Leg Raising; Diagnostic Test: Vena Cava Ultrasound; Diagnostic Test: End-expiratory /-inspiratory occlusion test; Drug: Fluid bolus

INTERVENTIONS:
Device: Transthoracic Echocardiography — Transthoracic echocardiography (TTE) is used for intermittent non-invasive stroke volume (SV) measurements. It is calculated by multiplication of left ventricular out flow tract (LVOT) and LVOT velocity time integral (VTI), obtained in a parasternal long axis view and apical five chamber view, respectively.
Device: Uncalibrated Pulse Contour Analysis — Pulse Contour Analysis allows an automated and continuous measurement of stroke volume (SV). Its underlying principle is that the integral of the systolic arterial pressure curve directly correlates with stroke volume.
Device: Transpulmonary Thermodilution/Calibrated Pulse Contour Analysis — Transpulmonary thermodilution (TPTD) involves the administration of a cold saline bolus into a central venous catheter. A special thermistor catheter placed in the femoral or brachial artery detects the successive changes in blood temperature. The resulting heat dissipation curve is analyzed to estimate stroke volume, cardiac output and other hemodynamic variables such as intrathoracic thermal volume (ITTV), pulmonary thermal volume (PTV), global end-diastolic volume (GEDV), intrathoracic blood volume (ITBV) and extravascular lung water (EVLW). Intermittent TPTD-derived cardiac output measurements (typically performed 1-3x/d) are used to calibrate pulse contour analysis.
Device: Esophageal Doppler — In esophageal Doppler, a thin ultrasound probe, coated with aqueous ultrasound gel, is orally or nasally inserted into the esophagus and orientated towards the aorta. By emission and detection of continuous wave Doppler signals, real time spectral waveforms of red blood cell velocity in the aorta are obtained, from which cardiac indices can be derived.
Device: Bioreactance — Bioreactance is a noninvasive hemodynamic monitoring technique, in which four double electrode sensors are placed on the skin of the chest. A high frequency sine wave is transmitted across the thorax. Pulsatile flow in the aorta causes phase shifts and amplitude changes of this signal, which are measured across the different electrodes and used to compute cardiac output.
Diagnostic Test: Passive Leg Raising — Passive Leg Raising (PLR) is a maneuver that mimics a fluid challenge by shifting about 300 ml of venous blood from the lower body to the heart. Thereby, it can help to predict fluid responsiveness without actual fluid infusion. To start with, the patient is placed in a semi-recumbent position. Then, the bed is adjusted so that the patient's torso is moved to a horizontal position and the lower limbs are raised to an angle of 45°. Hemodynamic effects occur and can be measured within one minute.
Diagnostic Test: Vena Cava Ultrasound — Inferior Vena Cava (IVC) Ultrasound has become a popular technique for assessing volume status. IVC diameter is measured in a subcostal long-axis IVC view 1-2 cm from the junction with the right atrium. The magnitude of distensibility during mechanical ventilation cycles or collapsibility during spontaneous breathing has been proposed to correlate with fluid responsiveness
Diagnostic Test: End-expiratory /-inspiratory occlusion test — In preload-dependent patients, mechanical ventilation induces periodic changes in cardiac output. Standardized maneuvers of end-expiratory or end-inspiratory interruption over 15 seconds may increase or decrease stroke volume, respectively, which is a valid predictor of fluid responsiveness
Drug: Fluid bolus — To verify fluid responsiveness, 500 ml of balanced crystalloids will be infused over a time of 15-20 min (25-33.33 ml/min) after completion of passive leg raising and restoration of baseline patient positioning

SUMMARY:
In extracorporeal membrane oxygenation (ECMO), blood is drawn out of the body via tubes, oxygenated in an artificial lung; and then pumped back into the blood vessels. This allows the supply of oxygen-rich blood to the organs (brain, heart, lungs, kidneys, liver, intestines, etc.) to be maintained. Continuous monitoring of cardiac function and circulatory status (blood pressure, blood flow to organs) is very important in intensive care medicine in order to control the administration of circulation-supporting medication and infusions. Various devices are routinely used for this task. However, in the specific situation of ECMO treatment, the measurements of these devices could be affected due to the artificial circulation; outside the body. The purpose of this study is therefore to test the accuracy of different methods of circulation monitoring during ECMO treatment.

DETAILED DESCRIPTION:
Hemodynamic monitoring and tests for fluid responsiveness are cornerstones of intensive care medicine. Generally, hemodynamic measurements can be obtained, for instance, with the following methods: pulmonary artery catheter, transthoracic echocardiography (TTE), esophageal doppler, transpulmonary thermodilution, pulse contour analysis and bioreactance, amongst others. Maneuvers for assessing volume responsiveness include passive leg raising (PLR), respiratory pulse pressure variation (PPV), stroke volume variation (SVV), inferior vena cava ultrasound (IVC), and end-inspiratory or end-expiratory occlusion tests. While these commonly used methods of hemodynamic assessment have been validated in various clinical scenarios, data are lacking in the setting of venoarterial extracorporeal membrane oxygenation (VA ECMO). VA ECMO is commonly used for circulatory support in patients with severe hemodynamic failure or cardiac arrest. Blood is most commonly drained from a femoral vein, pumped through an oxygenator, where it is oxygenated and decarboxylated, and thereafter reinfused into the patient via an arterial, most commonly femoral, return cannula. Theoretically, the artificial circulation with its blood drainage and return flows may interfere with common hemodynamic monitoring techniques and lead to erroneous measurements. The aim of this study therefore is to validate select techniques of hemodynamic monitoring and assessment of fluid responsiveness in patients on VA ECMO. In the context of this study, the performance of different hemodynamic monitoring tools and techniques for predicting fluid responsiveness will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patient receiving VA ECMO support
* Age 18 - 75 years

Exclusion Criteria:

* Pregnancy
* Conditions not allowing for passive leg raising maneuvers, e.g. "open abdomen", known or suspected elevation of intracranial pressure, recent leg or spinal trauma or orthopedic conditions not permitting leg raising
* Known ischemic or hemorrhagic stroke within 3 months prior to study enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Agreement of receiver operating characteristic (ROC) curves for predicting fluid responsiveness using the passive leg-raising test between different cardiac output measurement techniques (echocardiography, pulse contour analysis, thermodilution). | Repeated measurements throughout ECMO therapy (duration ranging from a few days to up to 24 weeks) and within up to 7 days after ECMO removal. Separate analysis for controlled and assisted mechanical ventilation.
  Cardiac Output (L/min) will be measured using transthoracic echocardiography, uncalibrated pulse contour analysis, and thermodilution before, during, and after a passive leg-raising test, as well as after administration of a fluid bolus of 500 ml balanced crystalloids over 15-20 min. A cardiac output increase of > 15% will be the cut-off for defining fluid responsiveness. Receiver operating characteristic (ROC) curves will be generated for each cardiac output measurement technique and compared using the Hanley-McNeil method. The agreement between the ROC curves (Hanley-McNeil test statistic) will serve as the primary outcome.

SECONDARY OUTCOMES:
Diagnostic performance (receiver operating characteristic (ROC) area under the curve) of an inspiratory and expiratory occlusion test in conjunction with pulse contour analysis for the prediction of fluid responsiveness during ECMO. | Repeated measurements throughout ECMO therapy (duration ranging from a few days to several weeks) and within a few days after ECMO removal. Separate analysis for controlled and assisted mechanical ventilation.
  Cardiac Output (L/min) will be measured using calibrated and uncalibrated pulse contour analysis before, during, and after an end-inspiratory and end-expiratory occlusion test (15 s), as well as after administration of a fluid bolus of 500 ml balanced crystalloids over 15-20 min. A cardiac output increase of > 15% after fluid infusion will be the cut-off for defining fluid responsiveness. Receiver operating characteristic (ROC) curves will be generated to assess the performance of the end-inspiratory and end-expiratory occlusion tests and the best threshold for predicting fluid responsiveness during ECMO.
Changes of cardiac output (L/min) over the course of ECMO therapy | Repeated measurements throughout ECMO therapy (duration ranging from a few days to up to 24 weeks) and within up to 7 days after ECMO removal.
  Cardiac output (L/min) will be measured at different time points (at least at the beginning of ECMO therapy and after ECMO removal) throughout ECMO therapy using transthoracic echocardiography, uncalibrated pulse contour analysis, and thermodilution.
Changes of tricuspid annular plane systolic excursion (TAPSE, mm) over the course of ECMO therapy | Repeated measurements throughout ECMO therapy (duration ranging from a few days to up to 24 weeks) and within up to 7 days after ECMO removal.
  Tricuspid annular plane systolic excursion (TAPSE, mm) will be measured at different time points (at least at the beginning of ECMO therapy and after ECMO removal) throughout ECMO therapy using transthoracic echocardiography.
Changes of tissue doppler imaging tricuspid annular velocity (cm/s) over the course of ECMO therapy | Repeated measurements throughout ECMO therapy (duration ranging from a few days to up to 24 weeks) and within up to 7 days after ECMO removal.
  Tissue doppler imaging tricuspid annular velocity (cm/s) will be measured at different time points (at least at the beginning of ECMO therapy and after ECMO removal) throughout ECMO therapy using transthoracic echocardiography.
Changes in cardiac output (L/min, measured by transthoracic echocardiography, uncalibrated pulse contour analysis, thermodilution) at different ECMO blood flow rates | During the first (up to 7) days of VA ECMO therapy.
  During the first days of VA ECMO therapy, cardiac output (L/min) will be measured repeatedly at different ECMO blood flow rates (baseline blood flow, blood flow reduced by 1 l/min, return to baseline blood flow, blood flow increased by 1 l/min) using transthoracic echocardiography, uncalibrated pulse contour analysis, and thermodilution.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication may be provided to qualified researchers with academic interest in hemodynamic monitoring. Data or samples shared will be coded, with no PHI included.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
URL: https://github.com/bernhardnagler/hemodynamecmonitoring_datasharing